CLINICAL TRIAL: NCT05264129
Title: A Phase 4, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, and Efficacy of the Concomitant Use of Ubrogepant for the Acute Treatment of Migraine in Subjects Taking Atogepant for the Preventive Treatment of Episodic Migraine
Brief Title: Study to Assess Adverse Events When Ubrogepant Tablets in Combination With Atogepant Tablets Are Used to Treat Adult Participants With Migraine
Acronym: TANDEM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M23-072
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Episodic Migraine
Keywords: Episodic Migraine; Ubrogepant; Atogepant; QULIPTA; UBRELVY
MeSH Terms: interventions — atogepant; ubrogepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atogepant + Ubrogepant (Experimental): Participants will receive atogepant for 12 weeks followed by atogepant + ubrogepant for 12 weeks.
  Interventions: Drug: Atogepant; Drug: Ubrogepant

INTERVENTIONS:
Drug: Atogepant — Oral Tablet
  Other Names: QULIPTA
Drug: Ubrogepant — Oral Tablet
  Other Names: UBRELVY

SUMMARY:
Migraine is a neurological disease characterized by moderate or severe headache, associated with nausea, vomiting, and/or sensitivity to light and sound. This study will assess the safety and efficacy of the combination use of ubrogepant for the acute treatment of migraine headache in participants taking atogepant once daily for preventive treatment of migraine.

Ubrogepant is an approved drug for the acute treatment of migraine. Atogepant is an approved drug for the preventive treatment of migraine. Approximately 235 adult participants with EM will be enrolled in approximately 45 sites in the United States.

Participants will receive oral atogepant tablets once daily (QD) for 12 weeks followed by continued atogepant treatment with ubrogepant tablets taken as needed for the next 12 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* At least 1-year history of migraine with or without aura consistent with a diagnosis according to the International Classification of Headache Disorders (ICHD)-3, 2018.
* History of 4 to 14 migraine days per month on average in the 3 months prior to Screening (Visit 1) in the investigator's judgment.

Exclusion Criteria:

- Clinically significant hematologic, endocrine, cardiovascular, cerebrovascular, pulmonary, renal, hepatic, gastrointestinal, or neurologic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (37):
- United States (37):
  - Achieve Clinical Research, LLC /ID# 244912, Birmingham, Alabama
  - Xenoscience, Inc /ID# 243506, Phoenix, Arizona
  - Excell Research, Inc /ID# 242590, Oceanside, California
  - Neurological Research Institute /ID# 244161, Santa Monica, California
  - George J. Rederich M.D. Inc. /ID# 242589, Torrance, California
  - Diablo Clinical Research /ID# 242592, Walnut Creek, California
  - Westside Center for Clinical Research /ID# 243287, Jacksonville, Florida
  - Suncoast Clinical Research /ID# 242463, New Port Richey, Florida
  - Meridien Research /ID# 243508, Orlando, Florida
  - Accel Research Sites - St Petersburg Clinical Research Unit /ID# 243091, St. Petersburg, Florida
  - Meridian Clinical Research (Neurology) - Savannah /ID# 242689, Savannah, Georgia
  - Clinical Research Atlanta - Headlands LLC /ID# 242661, Stockbridge, Georgia
  - Allied Physicians - Fort Wayne Neurological Center /ID# 243511, Fort Wayne, Indiana
  - Pharmasite Research, Inc. /ID# 243505, Baltimore, Maryland
  - Medstar Georgetown Neurology /ID# 243289, Chevy Chase, Maryland
  - QUEST Research Institute /ID# 243284, Farmington Hills, Michigan
  - Clinvest Research LLC /ID# 242597, Springfield, Missouri
  - Princeton Center for Clinical Research /ID# 242652, Skillman, New Jersey
  - Bio Behavioral Health, Inc /ID# 242643, Toms River, New Jersey
  - Dent Neurosciences Research Center, Inc. /ID# 242641, Amherst, New York
  - Central New York Clinical Research /ID# 242593, Manlius, New York
  - Rochester Clinical Research /ID# 242470, New York, New York
  - PMG Research of Raleigh LLC /ID# 243286, Raleigh, North Carolina
  - CTI Clinical Trial and Consulting /ID# 242884, Cincinnati, Ohio
  - Aventiv Research Columbus /ID# 242462, Columbus, Ohio
  - The Orthopedic Foundation /ID# 243292, New Albany, Ohio
  - Summit Research Network /ID# 242467, Portland, Oregon
  - Abington Neurological Associates - Abington /ID# 243291, Abington, Pennsylvania
  - WR-ClinSearch /ID# 242640, Chattanooga, Tennessee
  - FutureSearch Trials of Neurology /ID# 242690, Austin, Texas
  - DiscoveResearch, Inc /ID# 242469, Bryan, Texas
  - FutureSearch Trials of Dallas, LP /ID# 242658, Dallas, Texas
  - Protenium Clinical Research /ID# 244067, Hurst, Texas
  - ClinPoint Trials /ID# 242660, Waxahachie, Texas
  - Advanced Research Institute - Ridgeline /ID# 242662, Ogden, Utah
  - Highland Clinical Research /ID# 245159, Salt Lake City, Utah
  - Core Clinical Research /ID# 244436, Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 263 participants were enrolled and included in the intent-to-treat (ITT) population; 1 participant withdrew consent before receiving study drug and therefore was not included in the demographics or any analyses.
Groups:
- Atogepant 60 mg (Period 1): Participants will receive atogepant 60 mg tablets orally once daily for 12 weeks (Day 1 to Week 12) in Period 1.
- Atogepant 60 mg + Ubrogepant 100 mg (Period 2): Participants will receive atogepant 60 mg tablets orally once daily and ubrogepant 100 mg tablets orally as needed for an additional 12 weeks (Week 12 to Week 24) in Period 2.
Period: Period 1 Atogepant (Day1 to Wk12)
Arm/Group | Atogepant 60 mg (Period 1) | Atogepant 60 mg + Ubrogepant 100 mg (Period 2)
Started | 262 (One participant was screened and initially signed the informed consent form, but the participant withdrew consent prematurely discontinuing from the study before receiving study drug.) | 0
Completed | 221 | 0
Not Completed | 41 | 0
Period: Period 2 Atogepant+Ubrogepant (Wk12-24)
Arm/Group | Atogepant 60 mg (Period 1) | Atogepant 60 mg + Ubrogepant 100 mg (Period 2)
Started | 0 | 218 (Three participants who completed Period 1 did not enter Period 2.)
Completed | 0 | 203
Not Completed | 0 | 15

BASELINE CHARACTERISTICS:
Population: Overall safety population included all participants who received at least 1 dose of study drug. 263 participants were enrolled, but one participant withdrew consent prematurely discontinuing from the study before receiving study drug.
Groups:
- All Subjects: Participants will receive atogepant 60 mg tablets orally once daily for 12 weeks (Day 1 to Week 12) in Period 1 then atogepant 60 mg tablets orally once daily and ubrogepant 100 mg tablets orally as needed for an additional 12 weeks (Week 12 to Week 24) in Period 2.
Arm/Group | All Subjects
Number analyzed (Participants) | 262
Age, Customized [Count of Participants; unit: Participants]
  Age Group: < 20 years | 0
  Age Group: 20 to 29 years | 43
  Age Group: 30 to 39 years | 60
  Age Group: 40 to 49 years | 71
  Age Group: 50 to 59 years | 53
  Age Group: 60 to 69 years | 33
  Age Group: ≥ 70 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 235
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 44
  White | 205
  More than one race | 4
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. A treatment-emergent adverse event (TEAE) is an AE that occurs or worsens after receiving investigational study drug.
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to approximately 28 weeks)
Population: Safety Population 1 (all subjects who received ≥ 1 dose of study drug during the open-label atogepant treatment period) and Safety Population 2 (all subjects who received ≥ 1 dose of study drug during the open-label atogepant + ubrogepant concomitant-use treatment period).
Measure: Count of Participants; unit: Participants
Arm/Group | Atogepant 60 mg (Period 1) | Atogepant 60 mg + Ubrogepant 100 mg (Period 2)
Number analyzed (Participants) | 262 | 218
Participants | 130 | 94

2. Primary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Laboratory Values as Assessed by the Investigator
Description: Clinical laboratory test values are considered PCS if they meet either the lower-limit or higher-limit PCS criteria defined in the categories below. Percentage of participants with PCS laboratory values are summarized for chemistry, hematology, and urinalysis. Only those categories where at least 1 person had a non-PCS value at Baseline and met the PCS criterion at least once during post-baseline are reported.
Time Frame: Up to approximately 28 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Atogepant 60 mg (Period 1) | Atogepant 60 mg + Ubrogepant 100 mg (Period 2)
Number analyzed (Participants) | 262 | 218
participants
  Erythrocytes, Hematology (10^12/L): < 0.9 * LLN: number analyzed (Participants) | 251 | 213
  Erythrocytes, Hematology (10^12/L): < 0.9 * LLN | 3 | 3
  Hematocrit (fraction of 1): < 0.9 * LLN: number analyzed (Participants) | 253 | 215
  Hematocrit (fraction of 1): < 0.9 * LLN | 5 | 2
  Hemoglobin (g/L): < 0.9 * LLN: number analyzed (Participants) | 249 | 212
  Hemoglobin (g/L): < 0.9 * LLN | 6 | 3
  Leukocytes, Hematology (10^9/L): < 0.9 * LLN: number analyzed (Participants) | 248 | 211
  Leukocytes, Hematology (10^9/L): < 0.9 * LLN | 3 | 7
  Lymphocytes (10^9/L): < 0.7 * LLN: number analyzed (Participants) | 253 | 215
  Lymphocytes (10^9/L): < 0.7 * LLN | 1 | 0
  Lymphocytes (10^9/L): > 1.3 * ULN: number analyzed (Participants) | 253 | 215
  Lymphocytes (10^9/L): > 1.3 * ULN | 0 | 1
  Neutrophils (10^9/L): < 0.7 * LLN: number analyzed (Participants) | 251 | 214
  Neutrophils (10^9/L): < 0.7 * LLN | 4 | 1
  Neutrophils (10^9/L): > 1.3 * ULN: number analyzed (Participants) | 251 | 214
  Neutrophils (10^9/L): > 1.3 * ULN | 4 | 1
  Platelets (10^9/L): < 0.5 * LLN: number analyzed (Participants) | 252 | 216
  Platelets (10^9/L): < 0.5 * LLN | 0 | 1
  Alanine Aminotransferase (U/L): ≥ 3.0 * ULN: number analyzed (Participants) | 256 | 217
  Alanine Aminotransferase (U/L): ≥ 3.0 * ULN | 3 | 0
  Aspartate Aminotransferase (U/L): ≥ 3.0 * ULN: number analyzed (Participants) | 256 | 217
  Aspartate Aminotransferase (U/L): ≥ 3.0 * ULN | 1 | 0
  Bicarbonate (mmol/L): < 0.9 * LLN: number analyzed (Participants) | 254 | 215
  Bicarbonate (mmol/L): < 0.9 * LLN | 5 | 2
  Bilirubin, Chemistry (µmol/L): ≥ 1.5 * ULN: number analyzed (Participants) | 255 | 216
  Bilirubin, Chemistry (µmol/L): ≥ 1.5 * ULN | 2 | 2
  Calcium (mmol/L): < 0.9 * LLN: number analyzed (Participants) | 256 | 217
  Calcium (mmol/L): < 0.9 * LLN | 1 | 0
  Creatine Kinase (U/L): > 2.0 * ULN: number analyzed (Participants) | 252 | 215
  Creatine Kinase (U/L): > 2.0 * ULN | 9 | 5
  Glucose, Chemistry (mmol/L): < 0.8 * LLN: number analyzed (Participants) | 254 | 215
  Glucose, Chemistry (mmol/L): < 0.8 * LLN | 2 | 2
  Glucose, Chemistry (mmol/L): > 2.0 * ULN: number analyzed (Participants) | 254 | 215
  Glucose, Chemistry (mmol/L): > 2.0 * ULN | 2 | 1
  Lactate Dehydrogenase (U/L): > 3.0 * ULN: number analyzed (Participants) | 256 | 217
  Lactate Dehydrogenase (U/L): > 3.0 * ULN | 1 | 0
  Phosphate (mmol/L): < 0.9 * LLN: number analyzed (Participants) | 254 | 215
  Phosphate (mmol/L): < 0.9 * LLN | 1 | 1
  Phosphate (mmol/L): > 1.1 * ULN: number analyzed (Participants) | 254 | 215
  Phosphate (mmol/L): > 1.1 * ULN | 3 | 0
  Potassium (mmol/L): < 0.9 * LLN: number analyzed (Participants) | 256 | 217
  Potassium (mmol/L): < 0.9 * LLN | 0 | 1
  Potassium (mmol/L): > 1.1 * ULN: number analyzed (Participants) | 256 | 217
  Potassium (mmol/L): > 1.1 * ULN | 5 | 4
  Protein, Chemistry (g/L): < 0.9 * LLN: number analyzed (Participants) | 254 | 217
  Protein, Chemistry (g/L): < 0.9 * LLN | 3 | 2
  Glucose, Urinalysis: At least 1+: number analyzed (Participants) | 251 | 214
  Glucose, Urinalysis: At least 1+ | 4 | 0
  Protein, Urinalysis: At least 1+: number analyzed (Participants) | 243 | 206
  Protein, Urinalysis: At least 1+ | 38 | 39

3. Primary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Electrocardiograms (ECGs) Findings as Assessed by the Investigator
Description: 12-lead ECGs were performed at select study visits. Only those categories where at least 1 person had a non-PCS value at Baseline and met the PCS criterion at least once during postbaseline are reported.
Time Frame: Up to approximately 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Atogepant 60 mg (Period 1) | Atogepant 60 mg + Ubrogepant 100 mg (Period 2)
Number analyzed (Participants) | 262 | 218
participants
  PR Interval (msec): ≥ 250: number analyzed (Participants) | 243 | 211
  PR Interval (msec): ≥ 250 | 0 | 0
  QRS Interval (msec): ≥ 150: number analyzed (Participants) | 243 | 212
  QRS Interval (msec): ≥ 150 | 0 | 1
  QTcB (msec): > 500: number analyzed (Participants) | 243 | 212
  QTcB (msec): > 500 | 0 | 0
  QTcB (msec): Increase of > 60: number analyzed (Participants) | 243 | 212
  QTcB (msec): Increase of > 60 | 0 | 0
  QTcF (msec): > 500: number analyzed (Participants) | 243 | 212
  QTcF (msec): > 500 | 0 | 0
  QTcF (msec): Increase of > 60: number analyzed (Participants) | 243 | 212
  QTcF (msec): Increase of > 60 | 0 | 0

4. Primary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Vital Sign Measurements as Assessed by the Investigator
Description: PCS postbaseline vital sign values are summarized for categories: systolic and diastolic blood pressures [sitting and standing], pulse rate [sitting and standing], respiratory rate, temperature, weight. Only those categories where at least 1 person had a non-PCS value at Baseline and met the PCS criterion at least once during postbaseline are reported.
Time Frame: Up to approximately 28 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Atogepant 60 mg (Period 1) | Atogepant 60 mg + Ubrogepant 100 mg (Period 2)
Number analyzed (Participants) | 262 | 218
participants
  Sitting Systolic Blood Pressure (mmHg): ≤ 90 and Decrease of ≥ 20: number analyzed (Participants) | 244 | 205
  Sitting Systolic Blood Pressure (mmHg): ≤ 90 and Decrease of ≥ 20 | 4 | 2
  Standing Systolic Blood Pressure (mmHg): ≥ 180 and Increase of ≥ 20: number analyzed (Participants) | 255 | 215
  Standing Systolic Blood Pressure (mmHg): ≥ 180 and Increase of ≥ 20 | 1 | 0
  Standing Systolic Blood Pressure (mmHg): ≤ 90 and Decrease of ≥ 20: number analyzed (Participants) | 255 | 215
  Standing Systolic Blood Pressure (mmHg): ≤ 90 and Decrease of ≥ 20 | 2 | 2
  Sitting Diastolic Blood Pressure (mmHg): ≥ 105 and Increase of ≥ 15: number analyzed (Participants) | 244 | 205
  Sitting Diastolic Blood Pressure (mmHg): ≥ 105 and Increase of ≥ 15 | 1 | 1
  Standing Diastolic Blood Pressure (mmHg): ≥ 105 and Increase of ≥ 15: number analyzed (Participants) | 255 | 215
  Standing Diastolic Blood Pressure (mmHg): ≥ 105 and Increase of ≥ 15 | 5 | 3
  Standing Diastolic Blood Pressure (mmHg): ≤ 50 and Decrease of ≥ 15: number analyzed (Participants) | 255 | 215
  Standing Diastolic Blood Pressure (mmHg): ≤ 50 and Decrease of ≥ 15 | 1 | 1
  Sitting Pulse Rate (bpm): ≥ 120 and Increase of ≥ 15: number analyzed (Participants) | 244 | 205
  Sitting Pulse Rate (bpm): ≥ 120 and Increase of ≥ 15 | 0 | 1
  Sitting Pulse Rate (bpm): ≤ 50 and Decrease of ≥ 15: number analyzed (Participants) | 244 | 205
  Sitting Pulse Rate (bpm): ≤ 50 and Decrease of ≥ 15 | 4 | 2
  Standing Pulse Rate (bpm): ≥ 120 and Increase of ≥ 15: number analyzed (Participants) | 255 | 215
  Standing Pulse Rate (bpm): ≥ 120 and Increase of ≥ 15 | 1 | 2
  Standing Pulse Rate (bpm): ≤ 50 and Decrease of ≥ 15: number analyzed (Participants) | 255 | 215
  Standing Pulse Rate (bpm): ≤ 50 and Decrease of ≥ 15 | 1 | 0
  Weight (kg): Increase of ≥ 7%: number analyzed (Participants) | 257 | 217
  Weight (kg): Increase of ≥ 7% | 5 | 7
  Weight (kg): Decrease of ≥ 7%: number analyzed (Participants) | 257 | 217
  Weight (kg): Decrease of ≥ 7% | 16 | 28
  Orthostatic Systolic Blood Pressure (mmHg): ≤ -20: number analyzed (Participants) | 242 | 203
  Orthostatic Systolic Blood Pressure (mmHg): ≤ -20 | 12 | 7
  Orthostatic Diastolic Blood Pressure (mmHg): ≤ -15: number analyzed (Participants) | 242 | 203
  Orthostatic Diastolic Blood Pressure (mmHg): ≤ -15 | 6 | 10
  Orthostatic Pulse Rate (bpm): ≥ 25: number analyzed (Participants) | 242 | 203
  Orthostatic Pulse Rate (bpm): ≥ 25 | 10 | 7

5. Primary Outcome: Number of Participants With Suicidal Ideation and Behaviour Using 5-Point Scale of Columbia-Suicide Severity Rating Scale (C-SSRS) During the Open-Label Treatment Period
Description: C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and suicidal behavior.
  Suicidal ideation is classified on a 5-item scale: 1 (wish to be dead), 2 (nonspecific active suicidal thoughts), 3 (active suicidal ideation with any methods [not plan] without intent to act), 4 (active suicidal ideation with some intent to act, without specific plan), and 5 (active suicidal ideation with specific plan and intent).
  Suicidal behavior is classified on a 5-item scale: 0 (no suicidal behavior), 1 (preparatory acts or behavior), 2 (aborted attempt), 3 (interrupted attempt), and 4 (actual attempt).
  More than 1 classification can be selected provided they represent separate episodes. Suicidal ideation: Minimum total score 1, maximum total score 5; higher total scores indicate more suicidal ideation. Suicidal behavior: Minimum total score 0, maximum total score 4; higher total scores indicate more suicidal behavior.
Time Frame: Week 1 to Week 12 for Safety Population 1; Week 12 to Week 24 for Safety Population 2
Population: Safety Population 1 consisted of all subjects who received at least 1 dose of study drug during the open-label atogepant treatment period as well as Safety Population 2 consisted of all subjects who went on to receive at least 1 dose of study drug during the open-label atogepant + ubrogepant concomitant-use treatment period.
  The one subject with positive suicidal behavior was erroneously reported in the questionnaire and had not had a positive suicidal behavior throughout the study.
Measure: Number; unit: participants
Arm/Group | Atogepant 60 mg (Period 1) | Atogepant 60 mg + Ubrogepant 100 mg (Period 2)
Number analyzed (Participants) | 262 | 218
participants
  Suicidal Ideation | 0 | 2
  Suicidal Behavior | 0 | 1

6. Primary Outcome: Number of Participants With Suicidal Ideation and Behaviour Using 5-Point Scale of Columbia-Suicide Severity Rating Scale (C-SSRS) During the 4-Week Safety Follow-Up Period
Description: as for outcome 5
Time Frame: From last dose of study drug to 4 weeks after last dose of study drug. Overall median time on atogepant treatment was 85 days.
Population: Safety Population 1 consisted of all subjects who received at least 1 dose of study drug during the open-label atogepant treatment period. The statistical analysis plan (SAP) does not include the Safety Population 2 (all subjects who received at least 1 dose of study drug in Period 2) subgroup analyses for this primary outcome measure.
Measure: Number; unit: participants
Arm/Group | Atogepant 60 mg (Period 1)
Number analyzed (Participants) | 262
participants
  Suicidal Ideation During Follow-Up Period | 1
  Suicidal Behavior During Follow-Up Period | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time of informed consent to the end of the study. The median time on follow-up was 75.5 days from Visit 1 (Week -1) through end of Period 1 and 206 days from baseline through end of Period 2.
Arm/Group | Atogepant 60 mg (Period 1) | Atogepant 60 mg + Ubrogepant 100 mg (Period 2)
All-Cause Mortality (participants affected / at risk) | 0/263 | 0/218
Serious Adverse Events (participants affected / at risk) | 1/263 | 1/218
Other Adverse Events (participants affected / at risk) | 66/263 | 15/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atogepant 60 mg (Period 1) (N=263) | Atogepant 60 mg + Ubrogepant 100 mg (Period 2) (N=218)
MYELOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
URETEROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atogepant 60 mg (Period 1) (N=263) | Atogepant 60 mg + Ubrogepant 100 mg (Period 2) (N=218)
CONSTIPATION (Gastrointestinal disorders) | 14 (14) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 16 (16) | 2 (2)
FATIGUE (General disorders) | 17 (17) | 3 (3)
COVID-19 (Infections and infestations) | 23 (24) | 7 (7)
DECREASED APPETITE (Metabolism and nutrition disorders) | 15 (15) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT05264129/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT05264129/SAP_001.pdf